CLINICAL TRIAL: NCT06962384
Title: Comparative Analysis of Posterior Release Sclerotomy vs Conventional Ball Implantation in Evisceration Surgery
Brief Title: Comparing Posterior Release Sclerotomy With Conventional Evisceration Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Khaled Kotb Abdallah, Lecturer of ophthalmology fayoum university, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUH
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Evisceration; Ocular Trauma; Blind Painful Eye; Phthisis Bulbi; End Stage Glaucoma
Keywords: Evisceration; Ball implantation; Posterior release sclerotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posterior Release Sclerotomy Group (PRS Group) (Experimental): A key advancement in evisceration techniques is posterior release sclerotomy within the scleral cup, which aims to expand the intraocular space and facilitate primary ball implantation. By creating a controlled posterior opening, this method is hypothesized to reduce intraoperative resistance to implant insertion, minimize excessive intraocular pressure, and decrease postoperative complications such as extrusion or exposure
  Interventions: Procedure: Posterior release sclerotomy
- Conventional Ball Implantation Group (CBI Group) (Experimental): Conventional evisceration techniques involve creating a scleral incision to accommodate the ball implant, often requiring significant manipulation to fit the prosthesis securely. The resultant tight fit can lead to ischemic changes, delayed healing, and an increased risk of implant extrusion.
  Interventions: Procedure: Conventional Ball Implantation

INTERVENTIONS:
Procedure: Posterior release sclerotomy — * A 360-degree radial scleral incision was made, and an evisceration spoon was used to remove intraocular contents.
  * The scleral shell was cauterized to eliminate any residual uveal tissue.
  * Any remaining necrotic or inflamed tissue was debrided to ensure a clean surgical field and minimize postoperative complications.
  Posterior Release Sclerotomy Group (PRS Group)
  * A posterior sclerotomy (2-3 mm) was created at the posterior pole of the scleral shell using a crescent blade.
  * This sclerotomy expanded the intraocular space, reducing intraoperative resistance during implant insertion.
  * The spherical implant was gently placed within the expanded scleral shell, ensuring minimal stress on the tissue.
  Arms: Posterior Release Sclerotomy Group (PRS Group)
Procedure: Conventional Ball Implantation — * A 360-degree radial scleral incision was made, and an evisceration spoon was used to remove intraocular contents.
  * The scleral shell was cauterized to eliminate any residual uveal tissue.
  * Any remaining necrotic or inflamed tissue was debrided to ensure a clean surgical field and minimize postoperative complications.
  * No posterior sclerotomy was performed.
  * The implant was inserted directly into the scleral cup, requiring greater force to accommodate the implant within the available space.
  Arms: Conventional Ball Implantation Group (CBI Group)

SUMMARY:
The primary objective of this interventional study is to compare posterior release sclerotomy in the scleral cup with conventional ball implantation during evisceration, focusing on intraoperative feasibility, postoperative outcomes, and implant stability.

Specific objectives include:

1. Assessing the rate of implant migration and extrusion.
2. Evaluating the long-term stability of the implant within the scleral shell.
3. Investigating the occurrence of complications such as exposure or infection.
4. Analyzing the functional and anatomical outcomes.
5. Comparing patient satisfaction and quality of life measures.

DETAILED DESCRIPTION:
Evisceration is a widely performed ocular procedure aimed at removing intraocular contents while preserving the scleral shell and extraocular muscles. The primary goal of evisceration is to provide a structurally stable orbital implant, ensuring optimal prosthetic motility and cosmetic appearance. Traditional evisceration with ball implantation often presents complications related to limited space within the scleral cavity, potentially leading to implant extrusion or migration.

A key advancement in evisceration techniques is posterior release sclerotomy within the scleral cup, which aims to expand the intraocular space and facilitate primary ball implantation. By creating a controlled posterior opening, this method is hypothesized to reduce intraoperative resistance to implant insertion, minimize excessive intraocular pressure, and decrease postoperative complications such as extrusion or exposure. However, comparative studies on the effectiveness of posterior release sclerotomy versus conventional ball implantation remain limited.

Conventional evisceration techniques involve creating a scleral incision to accommodate the ball implant, often requiring significant manipulation to fit the prosthesis securely. The resultant tight fit can lead to ischemic changes, delayed healing, and an increased risk of implant extrusion. In contrast, posterior release sclerotomy allows for better distribution of intraocular pressure and improved accommodation of the implant, potentially reducing postoperative complications.

Several studies have highlighted the importance of scleral integrity and orbital volume restoration in optimizing prosthetic movement and overall aesthetic outcomes. Ensuring adequate implant placement without undue pressure on the scleral shell is a crucial factor in preventing long-term complications such as conjunctival dehiscence or implant migration. Posterior release sclerotomy may offer a surgical advantage by providing additional space for implantation, reducing undue pressure, and preserving the scleral integrity.

Despite these theoretical advantages, clinical evidence comparing posterior release sclerotomy with conventional ball implantation remains scarce. Previous retrospective studies suggest that modified techniques may enhance surgical ease and reduce complications.

The present study aims to compare posterior release sclerotomy in the scleral cup with conventional ball implantation during evisceration, focusing on intraoperative feasibility, postoperative outcomes, and implant stability.

This prospective, randomized, controlled trial will be conducted at the Department of Ophthalmic Surgery, Factuality of medicine, Fayum university.

The study will enroll patients requiring evisceration to one of two groups:

* Posterior Release Sclerotomy Group (PRS Group): Underwent evisceration with posterior release sclerotomy before primary ball implantation.
* Conventional Ball Implantation Group (CBI Group): Underwent standard evisceration with direct ball implantation without posterior sclerotomy.

  1. History Taking
* Ocular History: Duration and cause of blindness, previous surgeries/trauma, pain, inflammation, or medication use.
* Systemic History: Comorbidities (diabetes, hypertension, autoimmune diseases), history of radiation or malignancies.
* Medication History: Use of anticoagulants or immunosuppressants affecting bleeding or healing.

  2. Clinical Examination
* Visual Acuity Testing (if applicable)
* Slit-lamp Examination: Corneal clarity, conjunctival health, intraocular inflammation.
* Tonometry: Intraocular pressure measurement.
* Fundus Examination: To rule out intraocular pathology.
* External Examination: Eyelid position, orbital contour, tenderness, masses. 3. Preoperative Investigations
* CBC, Coagulation Profile .
* FBS & HbA1c.
* Orbital Ultrasound (if needed) : Assess scleral integrity.
* CT Orbit (if indicated): For suspected fractures, tumors.

Surgical Procedure All surgeries were performed under general anesthesia by an experienced ophthalmic surgeon. Standard sterile techniques were followed, and appropriate antibiotic prophylaxis was administered preoperatively.

1. Preoperative Preparation

   * Antibiotic prophylaxis: Intravenous cefazolin (1g) was given 30 minutes before surgery.
   * The surgical site was prepared with povidone-iodine 5%, and a lid speculum was placed.
   * A 360-degree conjunctival peritomy was performed using Westcott scissors, followed by meticulous dissection to expose the scleral shell.
2. Evisceration Procedure
3. Group-Specific Implantation Procedures Posterior Release Sclerotomy Group (PRS Group) Conventional Ball Implantation Group (CBI Group)

   * No posterior sclerotomy was performed.
   * The implant was inserted directly into the scleral cup, requiring greater force to accommodate the implant within the available space.
4. Closure and Conformer Placement

   * The scleral flaps were sutured in a purse-string fashion using non-absorbable 6-0 sutures.
   * The conjunctiva was closed with interrupted 8-0 Vicryl sutures to ensure proper healing.
   * A temporary conformer was placed inside the orbit to maintain the fornices and prevent conjunctival contracture.
   * The surgical site was padded and bandaged to provide adequate protection and minimize postoperative swelling.
5. Postoperative Care

   * Patients were monitored for early complications (e.g., bleeding, infection).
   * Topical antibiotics and corticosteroids were prescribed postoperatively.
   * Patients were followed up at 1 week, 1 month, and 6 months to assess implant stability, healing, and cosmetic outcomes.

Outcome Measures Primary Outcome

* Implant extrusion/migration rate within 6 months Secondary Outcomes
* Surgical ease and intraoperative difficulty score
* Postoperative pain (Visual Analogue Scale score)
* Healing time (conjunctival re-epithelialization)
* Implant stability and motility
* Cosmetic outcome (patient satisfaction scores, prosthesis motility)

Ethical consideration:

All the individuals included in the study will be informed about the procedures regarding the study and will be informed of their rights to refuse participation or withdraw from the study without having to give reasons. Participants will be guaranteed anonymity and all information provided would be treated with confidentiality. The ethical approval of the faculty of medicine, fayoum university research ethical committee (REC) will be obtained prior to the beginning of the work.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Indication for evisceration due to a non-malignant cause, such as painful blind eye, severe ocular trauma, end-stage glaucoma, or phthisis bulbi
* Adequate scleral integrity to allow for ball implantation
* No history of previous intraocular surgery or scleral weakening disorders

Exclusion Criteria:

* Orbital malignancy or suspected intraocular tumor
* Active ocular or periocular infection
* History of radiation therapy to the orbit
* Severe scleral thinning that contraindicates scleral preservation
* Presence of autoimmune disease affecting wound healing
* Psychiatric disorders affecting compliance with postoperative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
• Implant extrusion/migration rate within 6 months | Through study completion, an average of 6 months
  The primary outcome measure was implant stability, assessed clinically and through imaging at 1, 3, and 6 months postoperatively to review any signs of implant migration or extrusion as well as signs of conjunctival erosion.

SECONDARY OUTCOMES:
Patient satisfaction with implant motility | From enrollment to the end of the follow up period after 6 months
  Assessed through a standardized questionnaire. Measuring patient satisfaction by giving a score from 1-5, where 5 means excellent and 1 means very poor.
Postoperative pain | From enrollment to the end of the follow up period after 6 months
  The Quality of Life Score was determined using a Visual Analog Scale (VAS), which is a straight horizontal line, usually 10 mm. The ends of which are described as the extreme limits of the parameter to be measured oriented from the left (worst) to the right (best).
Postoperative complications | From enrollment to the end of the follow up period after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No